CLINICAL TRIAL: NCT00466180
Title: Adherence, Efficacy and Tolerance of Once-a-day Nevirapine-based Regimen in HIV-1 Infected Patients
Acronym: POSOVIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POSOVIR
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infections
Keywords: Once-a-day; Adherence; Nevirapine; Patient noncompliance; Administration and dosage; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Nevirapine from twice-a-day to once-a-day

SUMMARY:
Taking antiretrovirals once-a-day is considered the simpler way to improve adherence. However, it is not know if this assertion apply to patients taking their medication twice-a-day who change to once-a-day.

We hypothesized that once-daily dosing improves adherence.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults receiving antiretroviral therapy including nevirapine twice-a-day for at least 6 months
* plasma HIV RNA<400 cp/ml during the previous 4 months on 2 occasions
* accept adherence electronic monitoring
* written informed consent signed

Exclusion Criteria:

* asparate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5N if hepatitis virus B or C were negative
* AST or ALT>1.25N if hepatitis virus B or C were positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
MEMS adherence by electronic devices | 28-week period (randomized phase)

SECONDARY OUTCOMES:
Virologic efficacy (RNA HIV<400cp/ml)
Immunologic efficacy (CD4 count cells)
Tolerance (hepatic, cutaneous, ANRS safety grade scale)
Pharmacokinetics (nevirapine dosages)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Parienti, MD, Principal Investigator — University Hospital, Caen

REFERENCES:
- [Background] Parienti JJ, Das-Douglas M, Massari V, Guzman D, Deeks SG, Verdon R, Bangsberg DR. Not all missed doses are the same: sustained NNRTI treatment interruptions predict HIV rebound at low-to-moderate adherence levels. PLoS One. 2008 Jul 30;3(7):e2783. doi: 10.1371/journal.pone.0002783. PMID 18665246
- [Result] Parienti JJ, Massari V, Reliquet V, Chaillot F, Le Moal G, Arvieux C, Vabret A, Verdon R; POSOVIR Study Group. Effect of twice-daily nevirapine on adherence in HIV-1-infected patients: a randomized controlled study. AIDS. 2007 Oct 18;21(16):2217-22. doi: 10.1097/QAD.0b013e3282eff388. PMID 18090049